CLINICAL TRIAL: NCT00256386
Title: LabAlert: Enhancing Medication Safety Through Electronic Interventions to Improve Medication Safety
Brief Title: LabAlert: Enhancing Medication Safety Through Electronic Interventions to Improve Laboratory Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Garfield Memorial Fund (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 101-9520 Garfield Mem Trust
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2005-11

CONDITIONS: Safety
Keywords: Baseline; Laboratory; Drug
MeSH Terms: interventions — Electronic Health Records; Radiotherapy

INTERVENTIONS:
Device: Electronic Medical Record (EMR) to clinician's in-basket
Device: Automated Voice Message (AVM) reminder to patient's phone
Procedure: Pharmacy Team phone call-letter followup

SUMMARY:
Errors and preventable adverse events associated with medication prescription and dispensing are common, and the difference between guideline recommendations and the actual frequency of laboratory monitoring is substantial. This study evaluates three interventions to improve laboratory monitoring at initiation of medication therapy: an electronic medical record reminder to the prescribing clinician (EMR), an automated voice message to the patient (AVM), and a pharmacy team outreach (Pharmacy) compared to usual care (UC).

DETAILED DESCRIPTION:
Many of the medications that clinicians prescribe to prevent or treat disease can result in unanticipated and unintended toxic effects. Many national clinical guidelines recommend baseline and periodic laboratory monitoring to avoid adverse drug events. Our Safety in Prescribing project (SIP) has found many significant gaps in medication safety. Lab Alert will evaluate electronic tools to improve Kaiser Permanente's performance in laboratory monitoring to avoid adverse drug events. We will enroll patients who are taking high-risk medications and who have not received laboratory monitoring. The primary outcome of this 2-year study is the proportion of patients who receive guideline-based laboratory monitoring at 1 and 3 weeks post-intervention.

Fifteen primary care clinics will be randomly assigned to: (1) usual care (UC) (2) electronic message reminder (EMR) (3) automated voice message (AVM) (4) pharmacy outreach team (Pharmacy). The reminders will notify of the patient's need for guideline-specified laboratory testing due to medication use. Using electronic data, patients with PCPs assigned to intervention clinics who are on study-specified medications will be identified and screened for exclusions, to yield 600 patients (200 per intervention group). Patients will be assigned to the treatment groups on the basis of the condition assigned to their usual clinic. After the intervention and observation periods, and using the same time frame and inclusion and exclusion criteria used to identify the patients in the intervention arms, we will retrospectively identify a comparison 200-patient cohort in the usual care clinics. Thus, approximately 800 patients will be included in the study. Baseline, follow-up, and outcome data will be obtained from electronic records.

Study-defined medications will be finalized by the study team and quality committees. These medications are identified based upon previous work and are prescribed with reasonable frequency, commonly have gaps in laboratory monitoring, carry significant risk of toxicity, and are of interest to the participating HMOs because of prior and potential adverse events. We anticipate focusing on baseline monitoring for new prescriptions. New starts will be defined as patients with an index prescription but no other dispense of that medication in the prior 6 months.

Lab Alert will assess the effectiveness of a patient-specific electronic medical record (EMR) in-basket reminder to the primary care provider (PCP) (EMR reminder), an automated recorded voice message to the patient (AVM), pharmacy team outreach (Pharmacy) to increase the proportion of patients receiving all guideline-based laboratory monitoring, when compared to usual care (UC). If any intervention is better than UC, Lab Alert will assess and compare their effectiveness and costs. The study also will evaluate PCP and patient experiences with the intervention in order to refine the interventions in the future.

ELIGIBILITY:
Inclusion Criteria:

* Dispensed one of 12 drugs or classes of drugs where baseline safety laboratory monitoring is recommended and labs have not been completed 6 months prior or 5 days after the dispense of the medication.
* 18 years of age or older
* 12-month HMO membership
* drug benefit coverage
* has telephone number

Exclusion Criteria:

* recommended baseline laboratory monitoring completed
* receives care and/or resides in hospice, nursing home, care outside HMO
* enrolled in other care management program
* nonEnglish speaking needing translation services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2004-01; Study Completion 2005-03

PRIMARY OUTCOMES:
The number of patients that complete recommended laboratory monitoring within one week and twenty five days after intervention.
The study will evaluate the time to completion of the recommended labs.
The study will also evaluate PCP and patient experiences with the interventions in order to refine the interventions in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Adrianne C. Feldstein, MD, MS, Principal Investigator — Northwest Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Background] Brennan TA, Leape LL, Laird NM, Hebert L, Localio AR, Lawthers AG, Newhouse JP, Weiler PC, Hiatt HH. Incidence of adverse events and negligence in hospitalized patients. Results of the Harvard Medical Practice Study I. N Engl J Med. 1991 Feb 7;324(6):370-6. doi: 10.1056/NEJM199102073240604. PMID 1987460
- [Background] Beard K. Adverse reactions as a cause of hospital admission in the aged. Drugs Aging. 1992 Jul-Aug;2(4):356-67. doi: 10.2165/00002512-199202040-00008. PMID 1504448
- [Background] Classen DC, Pestotnik SL, Evans RS, Lloyd JF, Burke JP. Adverse drug events in hospitalized patients. Excess length of stay, extra costs, and attributable mortality. JAMA. 1997 Jan 22-29;277(4):301-6. PMID 9002492
- [Background] Burnum JF. Letter: Preventability of adverse drug reactions. Ann Intern Med. 1976 Jul;85(1):80-1. doi: 10.7326/0003-4819-85-1-80. No abstract available. PMID 937927
- [Background] Leape LL, Brennan TA, Laird N, Lawthers AG, Localio AR, Barnes BA, Hebert L, Newhouse JP, Weiler PC, Hiatt H. The nature of adverse events in hospitalized patients. Results of the Harvard Medical Practice Study II. N Engl J Med. 1991 Feb 7;324(6):377-84. doi: 10.1056/NEJM199102073240605. PMID 1824793
- [Background] Bates DW, Cullen DJ, Laird N, Petersen LA, Small SD, Servi D, Laffel G, Sweitzer BJ, Shea BF, Hallisey R, et al. Incidence of adverse drug events and potential adverse drug events. Implications for prevention. ADE Prevention Study Group. JAMA. 1995 Jul 5;274(1):29-34. PMID 7791255
- [Background] Thomas EJ, Studdert DM, Burstin HR, Orav EJ, Zeena T, Williams EJ, Howard KM, Weiler PC, Brennan TA. Incidence and types of adverse events and negligent care in Utah and Colorado. Med Care. 2000 Mar;38(3):261-71. doi: 10.1097/00005650-200003000-00003. PMID 10718351
- [Background] Gandhi TK, Burstin HR, Cook EF, Puopolo AL, Haas JS, Brennan TA, Bates DW. Drug complications in outpatients. J Gen Intern Med. 2000 Mar;15(3):149-54. doi: 10.1046/j.1525-1497.2000.04199.x. PMID 10718894
- [Background] Hulse RK, Clark SJ, Jackson JC, Warner HR, Gardner RM. Computerized medication monitoring system. Am J Hosp Pharm. 1976 Oct;33(10):1061-4. PMID 973633
- [Background] Lesar TS, Briceland L, Stein DS. Factors related to errors in medication prescribing. JAMA. 1997 Jan 22-29;277(4):312-7. PMID 9002494
- [Background] Graham DJ, Drinkard CR, Shatin D, Tsong Y, Burgess MJ. Liver enzyme monitoring in patients treated with troglitazone. JAMA. 2001 Aug 15;286(7):831-3. doi: 10.1001/jama.286.7.831. PMID 11497537
- [Background] Abookire SA, Karson AS, Fiskio J, Bates DW. Use and monitoring of
- [Background] Selby JV, Ettinger B, Swain BE, Brown JB. First 20 months' experience with use of metformin for type 2 diabetes in a large health maintenance organization. Diabetes Care. 1999 Jan;22(1):38-44. doi: 10.2337/diacare.22.1.38. PMID 10333901
- [Background] Beach JE, Faich GA, Bormel FG, Sasinowski FJ. Black box warnings in prescription drug labeling: results of a survey of 206 drugs. Food Drug Law J. 1998;53(3):403-11. No abstract available. PMID 10346718
- [Background] Raebel MA, Lyons EE, Andrade SE, Chan KA, Chester EA, Davis RL, Ellis JL, Feldstein A, Gunter MJ, Lafata JE, Long CL, Magid DJ, Selby JV, Simon SR, Platt R. Laboratory monitoring of drugs at initiation of therapy in ambulatory care. J Gen Intern Med. 2005 Dec;20(12):1120-6. doi: 10.1111/j.1525-1497.2005.0257.x. PMID 16423101
- [Background] Shea S, DuMouchel W, Bahamonde L. A meta-analysis of 16 randomized controlled trials to evaluate computer-based clinical reminder systems for preventive care in the ambulatory setting. J Am Med Inform Assoc. 1996 Nov-Dec;3(6):399-409. doi: 10.1136/jamia.1996.97084513. PMID 8930856
- [Background] Balas EA, Weingarten S, Garb CT, Blumenthal D, Boren SA, Brown GD. Improving preventive care by prompting physicians. Arch Intern Med. 2000 Feb 14;160(3):301-8. doi: 10.1001/archinte.160.3.301. PMID 10668831
- [Background] Rind DM, Safran C, Phillips RS, Wang Q, Calkins DR, Delbanco TL, Bleich HL, Slack WV. Effect of computer-based alerts on the treatment and outcomes of hospitalized patients. Arch Intern Med. 1994 Jul 11;154(13):1511-7. PMID 8018007
- [Background] Kaushal R, Shojania KG, Bates DW. Effects of computerized physician order entry and clinical decision support systems on medication safety: a systematic review. Arch Intern Med. 2003 Jun 23;163(12):1409-16. doi: 10.1001/archinte.163.12.1409. PMID 12824090
- [Background] Hoch I, Heymann AD, Kurman I, Valinsky LJ, Chodick G, Shalev V. Countrywide computer alerts to community physicians improve potassium testing in patients receiving diuretics. J Am Med Inform Assoc. 2003 Nov-Dec;10(6):541-6. doi: 10.1197/jamia.M1353. Epub 2003 Aug 4. PMID 12925546
- [Background] Freeborn DK PC. Promise and performance in managed care. Greenlick M, Freeborn D, Pope C, editors. 1994. Baltimore, MD, Johns Hopkins University Press.
- [Background] Feldstein AC, Smith DH, Robertson NR, Kovach CA, Soumerai SB, Simon SR, Sittig DF, Laferriere DS, Kalter M. Decision Support System Design and Implementation for Outpatient Prescribing: The Safety in Prescribing Study. In: Henriksen K, Battles JB, Marks ES, Lewin DI, editors. Advances in Patient Safety: From Research to Implementation (Volume 3: Implementation Issues). Rockville (MD): Agency for Healthcare Research and Quality (US); 2005 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK20567/ PMID 21250003
- [Background] Discount usability testing of computer-generated clinical alerts uncovers flaws. Denver, CO: 2003.
- [Background] Clark DO, Von Korff M, Saunders K, Baluch WM, Simon GE. A chronic disease score with empirically derived weights. Med Care. 1995 Aug;33(8):783-95. doi: 10.1097/00005650-199508000-00004. PMID 7637401
- [Background] Hosmer DWJr, Lemeshow S. Applied survival analysis: Regression modeling of time to event data. New York: Wiley and Sons, 1999.
- [Background] Raudenbush S, Bryk A, Cheong YF, Congdon R. HLM 5 hierarchical linear and nonlinear modeling. Lincolnwood: Scientific Software International, 2001.
- [Background] Schiff GD, Klass D, Peterson J, Shah G, Bates DW. Linking laboratory and pharmacy: opportunities for reducing errors and improving care. Arch Intern Med. 2003 Apr 28;163(8):893-900. doi: 10.1001/archinte.163.8.893. PMID 12719197
- [Background] Balas EA, Boren SA, Griffing G. Computerized management of diabetes: a synthesis of controlled trials. Proc AMIA Symp. 1998:295-9. PMID 9929229
- [Background] Bates DW. Using information technology to reduce rates of medication errors in hospitals. BMJ. 2000 Mar 18;320(7237):788-91. doi: 10.1136/bmj.320.7237.788. No abstract available. PMID 10720369
- [Background] Feldstein A, Elmer PJ, Smith DH, Herson M, Orwoll E, Chen C, Aickin M, Swain MC. Electronic medical record reminder improves osteoporosis management after a fracture: a randomized, controlled trial. J Am Geriatr Soc. 2006 Mar;54(3):450-7. doi: 10.1111/j.1532-5415.2005.00618.x. PMID 16551312
- [Background] Skipwith DH. Telephone counseling interventions with caregivers of elders. J Psychosoc Nurs Ment Health Serv. 1994 Mar;32(3):7-12. doi: 10.3928/0279-3695-19940301-05. PMID 8196022
- [Background] Poon EG, Gandhi TK, Sequist TD, Murff HJ, Karson AS, Bates DW.
- [Background] Smith CC, Bernstein LI, Davis RB, Rind DM, Shmerling RH. Screening for statin-related toxicity: the yield of transaminase and creatine kinase measurements in a primary care setting. Arch Intern Med. 2003 Mar 24;163(6):688-92. doi: 10.1001/archinte.163.6.688. PMID 12639201
- [Background] Krishna S, Balas EA, Boren SA, Maglaveras N. Patient acceptance of educational voice messages: a review of controlled clinical studies. Methods Inf Med. 2002;41(5):360-9. PMID 12501806
- [Background] Linkins RW, Dini EF, Watson G, Patriarca PA. A randomized trial of the effectiveness of computer-generated telephone messages in increasing immunization visits among preschool children. Arch Pediatr Adolesc Med. 1994 Sep;148(9):908-14. doi: 10.1001/archpedi.1994.02170090022002. PMID 8075732
- [Background] Leirer VO, Morrow DG, Pariante G, Doksum T. Increasing influenza vaccination adherence through voice mail. J Am Geriatr Soc. 1989 Dec;37(12):1147-50. doi: 10.1111/j.1532-5415.1989.tb06679.x. PMID 2592722
- [Background] Tanke ED, Leirer VO. Automated telephone reminders in tuberculosis care. Med Care. 1994 Apr;32(4):380-9. doi: 10.1097/00005650-199404000-00006. PMID 8139302
- [Background] Friedman RH, Kazis LE, Jette A, Smith MB, Stollerman J, Torgerson J, Carey K. A telecommunications system for monitoring and counseling patients with hypertension. Impact on medication adherence and blood pressure control. Am J Hypertens. 1996 Apr;9(4 Pt 1):285-92. doi: 10.1016/0895-7061(95)00353-3. PMID 8722429
- [Background] Friedman RH, Stollerman J, Rozenblyum L, Belfer D, Selim A, Mahoney D, Steinbach S. A telecommunications system to manage patients with chronic disease. Stud Health Technol Inform. 1998;52 Pt 2:1330-4. PMID 10384677
- [Background] Piette JD, Mah CA. The feasibility of automated voice messaging as an adjunct to diabetes outpatient care. Diabetes Care. 1997 Jan;20(1):15-21. doi: 10.2337/diacare.20.1.15. PMID 9028687
- [Background] Delichatsios HK, Friedman RH, Glanz K, Tennstedt S, Smigelski C, Pinto BM, Kelley H, Gillman MW. Randomized trial of a "talking computer" to improve adults' eating habits. Am J Health Promot. 2001 Mar-Apr;15(4):215-24. doi: 10.4278/0890-1171-15.4.215. PMID 11349340
- [Background] Raebel MA, Lyons EE, Chester EA, Bodily MA, Kelleher JA, Long CL, Miller C, Magid DJ. Improving laboratory monitoring at initiation of drug therapy in ambulatory care: a randomized trial. Arch Intern Med. 2005 Nov 14;165(20):2395-401. doi: 10.1001/archinte.165.20.2395. PMID 16287769
- [Background] Simon SR, Andrade SE, Ellis JL, Nelson WW, Gurwitz JH, Lafata JE, Davis RL, Feldstein A, Raebel MA. Baseline laboratory monitoring of cardiovascular medications in elderly health maintenance organization enrollees. J Am Geriatr Soc. 2005 Dec;53(12):2165-9. doi: 10.1111/j.1532-5415.2005.00498.x. PMID 16398903
- [Result] Feldstein AC, Smith DH, Perrin N, Yang X, Rix M, Raebel MA, Magid DJ, Simon SR, Soumerai SB. Improved therapeutic monitoring with several interventions: a randomized trial. Arch Intern Med. 2006 Sep 25;166(17):1848-54. doi: 10.1001/archinte.166.17.1848. PMID 17000941